CLINICAL TRIAL: NCT03251040
Title: Autologous Activated Fibrin Sealant for the Esophageal Anastomosis, a Feasibility Study
Brief Title: Fibrin Sealant in Esophageal Surgery
Acronym: SEAL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Responsible Party: Principal Investigator, Victor Plat, Principal investigator, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2015.458
Record Dates: First submitted 2017-08-07; First posted 2017-08-16 (Actual); Last update posted 2017-08-22 (Actual); Status verified 2017-08

CONDITIONS: Anastomotic Leak
Keywords: Esophagogastric anastomosis; Fibrin sealant; Sealing
MeSH Terms: conditions — Anastomotic Leak

STUDY DESIGN:
Intervention Model Description: Pilot study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fibrin sealant (Other): Single arm pilot study
  Interventions: Device: Autologous activated fibrin sealant

INTERVENTIONS:
Device: Autologous activated fibrin sealant — Application of fibrin sealant

SUMMARY:
Anastomotic leakage remains a major complication after esophageal surgery. Amongst other preventive measures, fibrin sealant is a promising adjunct to conventional anastomotic techniques. The investigators aimed to investigate feasibility of additional sealing by means of autologous fibrin sealant of the esophageal anastomosis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 - 90 years
* Scheduled to undergo elective minimal invasive esophageal surgery with thoracic or cervical anastomosis (i.e. Ivor Lewis, Orringer or McKeown esophagectomy).
* physical status (American Society of Anesthesiologists) of 3 or lower

Exclusion Criteria:

* Other malignancies
* Previous esophageal surgery were excluded

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-08-01 (Actual); Primary Completion 2016-04-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Anastomotic leakage | 30-day morbidity

CONTACTS AND LOCATIONS:
Overall Officials: Freek Daams, MD PhD, Study Director — Amsterdam UMC, location VUmc

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Plat VD, Bootsma BT, van der Wielen N, van der Peet DL, Daams F. Autologous Activated Fibrin Sealant for the Esophageal Anastomosis: A Feasibility Study. J Surg Res. 2019 Feb;234:49-53. doi: 10.1016/j.jss.2018.08.049. Epub 2018 Sep 27. PMID 30527497